CLINICAL TRIAL: NCT00742339
Title: Terlipressin + Albumin Versus Midodrine + Octreotide in the Treatment of Hepatorenal Syndrome (HRS): An Open Multicentric Randomized Study
Brief Title: Terlipressin + Albumin Versus Midodrine + Octreotide in the Treatment of Hepatorenal Syndrome
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Decision of independent monitoring committee: Risk of non-response to treatment significantly higher in midodrine group than in terlipressin group.
Sponsor: University of Padova (Other)
Responsible Party: Paolo Angeli, MD, PhD, Dept. of Clinical and Experimental Medicine, University of Padova, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1264P
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Cirrhosis; Hepatorenal Syndrome
Keywords: cirrhosis; hepatorenal syndrome; terlipressin; midodrine; octreotide; human albumin; effective circulating volume; The criteria which will be used for the diagnosis of HRS will be the criteria which were recently published by the International Ascites Club; Patients with cirrhosis and type 2 HRS only with serum creatinine value > 2.5 mg/dl; All patients with cirrhosis and type 1 HRS
MeSH Terms: conditions — Fibrosis; Hepatorenal Syndrome | interventions — Terlipressin; Albumins; Midodrine; Octreotide; Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Fifty patients with cirrhosis and HRS will be randomly assigned to arm 1.
  Interventions: Drug: Terlipressin plus albumin
- 2 (Experimental): Fifty patients with cirrhosis and HRS will be randomly assigned to arm 2.
  Interventions: Drug: Midodrine plus octreotide plus human albumin

INTERVENTIONS:
Drug: Terlipressin plus albumin — The terlipressin will be give at the initial dose of 3 mg/24 hours by intravenous continuous infusion. If during the following 48 hours the serum value of creatinine will not change or will go down less than 25%, the dose of terlipressin will be increased to 6 mg/24 hours. If no response will ensue, the dose of terlipressin will be increased to the maximal dose of 12 mg/24 hours. Twenty percent human albumin solution will be administrate together with terlipressin at the dosage of 1 g/Kg of body weight, on first day, and then, to the dosage of 20-40 g/Kg in order to maintain the central venous pressure (CVP) between 10 and 15 cm H2O.The treatment with terlipressin and albumin will be maintained for 24 hours after complete or incomplete resolution. The length of the study in patients with complete and incomplete resolution will reach a maximum of 15 days. In the patients without response the treatment with the high dosage of terlipressin will go on for a maximum of 7 days.
  Arms: 1
Drug: Midodrine plus octreotide plus human albumin — Midodrine will be give orally at the initial dose 7.5 tid together with octreotide at the initial dosage of 100 µg subcutaneously tid. If during the following 96 hours the serum value of creatinine will not change or will go down less than 25%, the dose of midodrine will be increased to 12.5 mg tid Twenty percent human albumin solution will be administrate together with midodrine and octreotide at the dosage of 1 g/Kg of body weight, on first day, and then, to the dosage of 20-40 g/Kg in order to maintain the central venous pressure (CVP) between 10 and 15 cm H2O.The treatment with terlipressin and albumin will be maintained for 24 hours after complete or incomplete resolution. The length of the study in patients with complete and incomplete resolution will reach a maximum of 15 days. In the patients without response the treatment with the high dosage of terlipressin will go on for a maximum of 7 days.
  Arms: 2

SUMMARY:
From 1999, several studies have showed that the use of vasoconstrictors in association with albumin are effective in the treatment of hepatorenal syndrome (HRS). The rationale of the use of vasoconstrictors together with albumin in the treatment of this severe complication of portal hypertension in patients with cirrhosis is to correct the reduction of the effective circulating volume due to the splanchnic arterial vasodilatation.In most of these studies terlipressin, a derivate of vasopressin, has been used as vasoconstrictor as intravenous boluses moving from an initial dose of 0.5-1 mg/4 hr. In some studies midodrine, an alpha-adrenergic agonist, given by mouth has been used as vasoconstrictor at a dose ranging from 2.5 up to 12.5 tid together with octreotide, an inhibitor of the release of glucagon, given subcutaneously at a dose ranging from 10 µg upt to 200 µg tid. To the day, there isn't a study comparing terlipressin + albumin versus midodrine + octreotide + albumin in the treatment of HRS in patients with cirrhosis.Thus, the aim of the study is to compare terlipressin + albumin vs midodrine + octreotide + albumin in the treatment of the HRS in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and diagnosis of HRS type 1 or 2,serum creatinine > 2.5 mg/dl

Exclusion Criteria:

* Diagnosis of HCC with a staging beyond the Milan Criteria di Milano
* Septic shock (systolic arterial pressure < 90 mmHg
* Significant heart or respiratory failure
* Peripheral arteriophaty clinically significant
* Previous heart stroke or significant alteration of the ECG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The primary end-point of the study is the complete reform of the renal function (serum creatinine < 1.5 mg/dl. The primary end point will be evaluated at the end of the treatment. | The treatment will be continued for a maximum of 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Clinical and Experimental Medicine, University of Padova, Padua, Italy

REFERENCES:
- [Background] Salerno F, Gerbes A, Gines P, Wong F, Arroyo V. Diagnosis, prevention and treatment of hepatorenal syndrome in cirrhosis. Gut. 2007 Sep;56(9):1310-8. doi: 10.1136/gut.2006.107789. Epub 2007 Mar 27. No abstract available. PMID 17389705